CLINICAL TRIAL: NCT01078545
Title: Lucrin® Depot Efficacy and Safety Monitoring Study in Patients With Advanced Prostate Cancer and Lower Urinary Tract Symptoms. International, Multicenter Post-marketing Observational Study.
Brief Title: Lucrin® Depot Efficacy and Safety Monitoring Study in Patients With Advanced Prostate Cancer and Lower Urinary Tract Symptoms (LUTS)
Acronym: LEMON
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Fraktal.com.pl (Unknown); Med-net.pl (Unknown)
Responsible Party: Sponsor
Other Study IDs: P10-612
Record Dates: First submitted 2010-02-28; First posted 2010-03-02 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Prostate Cancer; Lower Urinary Tract Symptoms
Keywords: Prostate cancer; Lower urinary tract symptoms; Hormonotherapy; LHRH analogue; Androgen deprivation therapy (ADT)
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adv. PCa patients with LUTS treated with GnRH analogue: Patients with advanced prostate cancer and lower urinary tract symptoms treated with GnRH analogue Lucrin Depot 11.25 mg (Lucrin Depot 3.75mg - in Ukraine)
  Interventions: Drug: Leuprolide acetate Depot Susp. 11.25 mg (Poland), 3.75 mg (Ukraine)

INTERVENTIONS:
Drug: Leuprolide acetate Depot Susp. 11.25 mg (Poland), 3.75 mg (Ukraine) — Leuprolide acetate 11.25 mg every 3 months sc or im, number of injections during the trial - 5 in Poland, Leuprolide acetate 3.75 mg every 1 month sc or im, number of injections during the trial - 12 in Ukraine.
  Other Names: Lupron Depot/Leuprolide acetate 11.25 mg; Lucrin Depot 11.25 mg; Lupron Depot/Leuprolide acetate 3.75 mg; Lucrin Depot 3.75 mg

SUMMARY:
The purpose of the study is to determine the influence of GnRH (gonadotropin releasing hormone) analogue - Lucrin Depot 11.25 mg (Lucrin Depot 3.75mg - in Ukraine) administration on intensity of lower urinary tract symptoms (LUTS) in patients with diagnosed locally advanced and/or metastatic prostate cancer and LUTS.

DETAILED DESCRIPTION:
The remaining target is:

- to assess the intensity of LUTS in Polish and Ukrainian patients with locally advanced and metastatic prostate cancer, previously untreated with hormonal therapy

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Locally advanced (T3-T4) and/or metastatic (N+/M+) hormone-sensitive prostate cancer, confirmed by histological examination
* Presence of lower urinary tract symptoms (LUTS)-IPSS >0
* Treatment with Lucrin® Depot is the routine therapy in the patient. The decision as to Lucrin® Depot choice will not be associated with patient's participation in the study, but will result from the best medical knowledge and practice.
* Until inclusion into PMOS the patient has not been treated with GnRH analogue.
* The patient, before inclusion into the study, has not been treated by surgery (radical prostatectomy).

Exclusion Criteria:

* Patients will not be included into the study if any contraindications to treatment with Lucrin® Depot exist, or if there are other treatment options which, according to the present medical knowledge, are potentially more beneficial for the patient.
* Physician or patient can stop treatment at any moment, if any indications or reasons exist.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Haczynski, MD, PhD, Study Director — Abbott Laboratories, Poland
Locations (143):
- Poland (132):
  - Site Reference ID/Investigator# 31076, Bełchatów
  - Site Reference ID/Investigator# 31002, Bialystok
  - Site Reference ID/Investigator# 30977, Bialystok
  - Site Reference ID/Investigator# 31030, Bialystok
  - Site Reference ID/Investigator# 31048, Bialystok
  - Site Reference ID/Investigator# 31083, Bobrowniki
  - Site Reference ID/Investigator# 31028, Bydgoszcz
  - Site Reference ID/Investigator# 31014, Bytom
  - Site Reference ID/Investigator# 31006, Bytom
  - Site Reference ID/Investigator# 31018, Bytom
  - Site Reference ID/Investigator# 31007, Ciechanów
  - Site Reference ID/Investigator# 31004, Elblag
  - Site Reference ID/Investigator# 31090, Elblag
  - Site Reference ID/Investigator# 31044, Ełk
  - Site Reference ID/Investigator# 30994, Florentynów
  - Site Reference ID/Investigator# 9803, Gdansk
  - Site Reference ID/Investigator# 31057, Gdansk
  - Site Reference ID/Investigator# 31101, Gdansk
  - Site Reference ID/Investigator# 31097, Gdansk
  - Site Reference ID/Investigator# 30984, Gliwice
  - Site Reference ID/Investigator# 30976, Gmina Brwinów
  - Site Reference ID/Investigator# 31009, Gmina Poddębice
  - Site Reference ID/Investigator# 31051, Imielnik Stary
  - Site Reference ID/Investigator# 31023, Inowrocław
  - Site Reference ID/Investigator# 31074, Inowrocław
  - Site Reference ID/Investigator# 31032, Jankowo
  - Site Reference ID/Investigator# 31067, Jarosławiec
  - Site Reference ID/Investigator# 30995, Jastków
  - Site Reference ID/Investigator# 31065, Jastrzębie Zdrój
  - Site Reference ID/Investigator# 31031, Jastrzębie Zdrój
  - Site Reference ID/Investigator# 31054, Jelenia Góra
  - Site Reference ID/Investigator# 30997, Katowice
  - Site Reference ID/Investigator# 31036, Katowice
  - Site Reference ID/Investigator# 31055, Kielce
  - Site Reference ID/Investigator# 30999, Kielce
  - Site Reference ID/Investigator# 31102, Kluczbork
  - Site Reference ID/Investigator# 31068, Kolbudy
  - Site Reference ID/Investigator# 31020, Konin
  - Site Reference ID/Investigator# 31019, Krakow
  - Site Reference ID/Investigator# 31087, Krakow
  - Site Reference ID/Investigator# 31050, Krakow
  - Site Reference ID/Investigator# 31025, Krakow
  - Site Reference ID/Investigator# 31043, Krakow
  - Site Reference ID/Investigator# 31011, Krakow
  - Site Reference ID/Investigator# 31061, Krakow
  - Site Reference ID/Investigator# 31053, Krakow
  - Site Reference ID/Investigator# 31029, Kurów
  - Site Reference ID/Investigator# 31012, Legnica
  - Site Reference ID/Investigator# 31040, Leszno
  - Site Reference ID/Investigator# 31082, Lidzbark Warmiński
  - Site Reference ID/Investigator# 31086, Lodz
  - Site Reference ID/Investigator# 31052, Lodz
  - Site Reference ID/Investigator# 31047, Lodz
  - Site Reference ID/Investigator# 31089, Lodz
  - Site Reference ID/Investigator# 31060, Lodz
  - Site Reference ID/Investigator# 31049, Lublin
  - Site Reference ID/Investigator# 31100, Lublin
  - Site Reference ID/Investigator# 33278, Lublin
  - Site Reference ID/Investigator# 31103, Lublin
  - Site Reference ID/Investigator# 31104, Lublin
  - Site Reference ID/Investigator# 30998, Lublin
  - Site Reference ID/Investigator# 31056, Michałowice
  - Site Reference ID/Investigator# 31001, Milcz
  - Site Reference ID/Investigator# 31085, Nysa
  - Site Reference ID/Investigator# 30993, Oborniki Śląskie
  - Site Reference ID/Investigator# 30974, Olsztyn
  - Site Reference ID/Investigator# 31080, Olsztyn
  - Site Reference ID/Investigator# 30989, Opole
  - Site Reference ID/Investigator# 30978, Opole
  - Site Reference ID/Investigator# 30982, Opole
  - Site Reference ID/Investigator# 31033, Opole
  - Site Reference ID/Investigator# 31075, Opole
  - Site Reference ID/Investigator# 31042, Ostrów Wielkopolski
  - Site Reference ID/Investigator# 31000, Piotrkow Trybunalski
  - Site Reference ID/Investigator# 31069, Piła
  - Site Reference ID/Investigator# 31045, Poznan
  - Site Reference ID/Investigator# 31088, Poznan
  - Site Reference ID/Investigator# 31021, Poznan
  - Site Reference ID/Investigator# 31058, Poznan
  - Site Reference ID/Investigator# 31034, Poznan
  - Site Reference ID/Investigator# 30985, Poznan
  - Site Reference ID/Investigator# 30979, Puszczykowo
  - Site Reference ID/Investigator# 31005, Puławy
  - Site Reference ID/Investigator# 31064, Puławy
  - Site Reference ID/Investigator# 31022, Pyskowice
  - Site Reference ID/Investigator# 31013, Płock
  - Site Reference ID/Investigator# 31016, Radlin
  - Site Reference ID/Investigator# 31099, Radom
  - Site Reference ID/Investigator# 31041, Rzeszów
  - Site Reference ID/Investigator# 31024, Siedlce
  - Site Reference ID/Investigator# 30988, Siemianowice Śląskie
  - Site Reference ID/Investigator# 31063, Sieradz
  - Site Reference ID/Investigator# 31015, Sosnowiec
  - Site Reference ID/Investigator# 30983, Starachowice
  - Site Reference ID/Investigator# 31084, Suwałki
  - Site Reference ID/Investigator# 31092, Suwałki
  - Site Reference ID/Investigator# 33277, Suwałki
  - Site Reference ID/Investigator# 31008, Swarzędz
  - Site Reference ID/Investigator# 30975, Szczecin
  - Site Reference ID/Investigator# 31046, Szczecin
  - Site Reference ID/Investigator# 30992, Szczecin
  - Site Reference ID/Investigator# 31035, Szczecin
  - Site Reference ID/Investigator# 31003, Świętochłowice
  - Site Reference ID/Investigator# 31079, Tarnowskie Góry
  - Site Reference ID/Investigator# 31071, Tarnów
  - Site Reference ID/Investigator# 31091, Tarnów
  - Site Reference ID/Investigator# 30980, Tomaszów Mazowiecki
  - Site Reference ID/Investigator# 31059, Torun
  - Site Reference ID/Investigator# 30987, Turek
  - Site Reference ID/Investigator# 31066, Warsaw
  - Site Reference ID/Investigator# 31037, Warsaw
  - Site Reference ID/Investigator# 31105, Warsaw
  - Site Reference ID/Investigator# 31106, Warsaw
  - Site Reference ID/Investigator# 31093, Warsaw
  - Site Reference ID/Investigator# 31094, Warsaw
  - Site Reference ID/Investigator# 31095, Warsaw
  - Site Reference ID/Investigator# 31081, Warsaw
  - Site Reference ID/Investigator# 31078, Warsaw
  - Site Reference ID/Investigator# 30986, Wieliczka
  - Site Reference ID/Investigator# 31027, Wroclaw
  - Site Reference ID/Investigator# 31038, Wroclaw
  - Site Reference ID/Investigator# 31062, Wroclaw
  - Site Reference ID/Investigator# 31070, Wroclaw
  - Site Reference ID/Investigator# 31077, Wroclaw
  - Site Reference ID/Investigator# 31072, Wroclaw
  - Site Reference ID/Investigator# 31098, Zabrze
  - Site Reference ID/Investigator# 30996, Zamość
  - Site Reference ID/Investigator# 31073, Złotniki
  - Site Reference ID/Investigator# 30981, Żory
  - Site Reference ID/Investigator# 31010, Łask
  - Site Reference ID/Investigator# 31096, Łazy
  - Site Reference ID/Investigator# 31039, Łomża
- Ukraine (11):
  - Site Reference ID/Investigator# 31108, Dnipro
  - Site Reference ID/Investigator# 31109, Dnipro
  - Site Reference ID/Investigator# 31111, Donetsk
  - Site Reference ID/Investigator# 31112, Kharkiv
  - Site Reference ID/Investigator# 31113, Kharkiv
  - Site Reference ID/Investigator# 31114, Kharkiv
  - Site Reference ID/Investigator# 31209, Kiev
  - Site Reference ID/Investigator# 31110, Kiev
  - Site Reference ID/Investigator# 21103, Kiev
  - Site Reference ID/Investigator# 31107, Kiev
  - Site Reference ID/Investigator# 31115, Simferopol

RESULTS

PARTICIPANT FLOW:
Groups:
- Advanced PCa Patients With LUTS Treated With GnRH Analogue: Patients with advanced prostate cancer (PCa) and lower urinary tract symptoms (LUTS) treated with GnRH analogue Lucrin Depot 11.25 mg (Lucrin Depot 3.75mg - in Ukraine)
Period: Overall Study
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Started | 729
Intent-to-treat Population | 729
Per Protocol Population | 661
Completed | 703
Not Completed | 26
Not completed — Lost to Follow-up | 13
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 3
Not completed — Death | 3
Not completed — Participant moved to another physician | 1

BASELINE CHARACTERISTICS:
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Number analyzed (Participants) | 729
Age Continuous [Mean (Standard Deviation); unit: years] | 71.2 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 729
Region of Enrollment [Number; unit: participants]
  Poland | 659
  Ukraine | 70
Age at diagnosis of prostate cancer [Mean (Standard Deviation); unit: years] — Age of participant when diagnosed with prostate cancer. Results based on 724 participants.
  years | 70.7 (7.1)
Prostate-Specific Antigen (PSA) concentration [Mean (Standard Deviation); unit: ng/mL] — The mean prostate-specific antigen (PSA) concentration at Baseline. Results based on 718 participants.
  ng/mL | 55.8 (291.5)
Prostate cancer type [Number; unit: Participants]
  Locally advanced | 562
  Advanced with metastases | 127
  Localized | 39
  Lack of data | 1
Gleason score [Number; unit: participants] — The Gleason score classifies each participant's prostate cancer based on how the cells look under the microscope. Prostate cancers often have areas with different grades, so a grade is assigned to the 2 areas that make up most of the cancer. The Gleason score is the sum of these 2 grades, resulting in a number from 2 to 10. The higher the Gleason score the more likely it is that the cancer will grow faster and spread beyond the prostate.
  participants
    2 | 1
    3 | 3
    4 | 35
    5 | 53
    6 | 151
    7 | 262
    8 | 167
    9 | 41
    10 | 13
    Lack of data | 3

OUTCOME MEASURES:

1. Primary Outcome: The Change in the International Prostate Symptom Score (IPSS) From Baseline to Month 12. The IPSS Has a Range From 0 to 35.
Description: The International Prostate Symptom Score (IPSS) is used to assess the severity of lower urinary tract symptoms (LUTS) and to monitor disease progression. The IPSS is calculated from 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, and straining [rated as 0 (not at all) to 5 (almost always)], as well as how many times on average a participant has to get up to urinate at night (0=none to 5=5 times or more). The total score is classified as follows: 0 to 7 = mildly symptomatic; 8 to 19 = moderately symptomatic; and 20 to 35 = severely symptomatic.
Time Frame: Baseline to 12 months
Population: Analysis conducted in the intent-to-treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Number analyzed (Participants) | 729
units on a scale
  IPSS at Baseline (n=727) | 17.8 (6.9)
  IPSS at 12 months (n=699) | 10.0 (5.0)

2. Secondary Outcome: The Change in the International Prostate Symptom Score (IPSS) From Baseline to 3, 6, 9, and 12 Months.
Description: as for outcome 1
Time Frame: Baseline to 3, 6, 9, and 12 months.
Population: Analysis conducted in the intent-to-treat population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Number analyzed (Participants) | 729
units on a scale
  IPSS at Baseline (n=727) | 17.8 (6.9)
  IPSS at month 3 (n=724) | 14.0 (5.6)
  IPSS at month 6 (n=717) | 12.3 (5.1)
  IPSS at month 9 (n=702) | 10.9 (4.9)
  IPSS at month 12 (n=699) | 10.0 (5.0)

3. Secondary Outcome: Percentage of Patients at Baseline With One of the Symptoms Connected With Prostate Cancer.
Description: Percentage of participants at baseline with one of the following symptoms connected with prostate cancer: hematospermia (blood in the sperm), lower abdominal pain, urine incontinence, erectile dysfunction, crotch pain, anal pain or bleeding, lumbar/back pain, bone pain, spinal compression symptoms, peripheral lymph node enlargement, and lymphatic oedema of lower extremities. The intensity of each symptom was rated by the participant from 1 (minimum) to 7 (maximum). Zero indicates that the symptom was not present.
Time Frame: Baseline
Population: Analysis conducted in the intent-to-treat population.
Measure: Number; unit: Percentage of participants
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Number analyzed (Participants) | 729
Percentage of participants
  Hematospermia | 3
  Lower abdominal pain | 31
  Urine incontinence | 13
  Erectile dysfunction | 62
  Crotch pain | 24
  Anal pain or bleeding | 2
  Lumbar/back pain | 15
  Bone pain | 17
  Spinal compression symptoms | 1
  Peripheral lymph node enlargement | 2
  Lymphatic oedema of the lower extremities | 6

4. Secondary Outcome: Changes in the Intensity of Symptoms Connected With Prostate Cancer From Baseline to Month 3, 6, 9, and 12.
Description: Changes in the intensity of the following symptoms connected with prostate cancer: hematospermia (blood in the sperm), lower abdominal pain, urine incontinence, erectile dysfunction, crotch pain, anal pain or bleeding, lumbar/back pain, bone pain, spinal compression symptoms, peripheral lymph node enlargement, and lymphatic oedema of lower extremities. The intensity of each symptom was rated by the participant from 1 (minimum) to 7 (maximum). Zero indicates that the symptom was not present.
Time Frame: Baseline to 3, 6, 9, and 12 months.
Population: Analysis conducted in the intent-to-treat population.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Number analyzed (Participants) | 729
Units on a scale
  Hematospermia (Baseline; n=729) | 0 [0 to 5]
  >Month 3 (n=726) | 0 [0 to 4]
  >Month 6 (n=719) | 0 [0 to 4]
  >Month 9 (n=704) | 0 [0 to 5]
  >Month 12 (n=703) | 0 [0 to 3]
  Lower abdominal pain (Baseline; n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 7]
  >Month 6 (n=719) | 0 [0 to 6]
  >Month 9 (n=704) | 0 [0 to 6]
  >Month 12 (n=703) | 0 [0 to 7]
  Urinary incontinence (Baseline; n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 7]
  >Month 6 (n=719) | 0 [0 to 7]
  >Month 9 (n=704) | 0 [0 to 7]
  >Month 12 (n=703) | 0 [0 to 7]
  Erectile dysfunction (Baseline; n=729) | 4 [0 to 7]
  >Month 3 (n=726) | 5 [0 to 7]
  >Month 6 (n=719) | 5 [0 to 7]
  >Month 9 (n=704) | 6 [0 to 7]
  >Month 12 (n=703) | 6 [0 to 7]
  Crotch pain (Baseline; n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 7]
  >Month 6 (n=719) | 0 [0 to 7]
  >Month 9 (n=704) | 0 [0 to 7]
  >Month 12 (n=703) | 0 [0 to 7]
  Anal pain or bleeding (Baseline; n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 7]
  >Month 6 (n=719) | 0 [0 to 4]
  >Month 9 (n=704) | 0 [0 to 4]
  >Month 12 (n=703) | 0 [0 to 3]
  Lumbar/back pain (Baseline n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 5]
  >Month 6 (n=719) | 0 [0 to 6]
  >Month 9 (n=704) | 0 [0 to 6]
  >Month 12 (n=703) | 0 [0 to 6]
  Bone pain (Baseline; n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 7]
  >Month 6 (n=719) | 0 [0 to 7]
  >Month 9 (n=704) | 0 [0 to 7]
  >Month 12 (n=703) | 0 [0 to 7]
  Spinal compression symptoms (Baseline; n=729) | 0 [0 to 5]
  >Month 3 (n=726) | 0 [0 to 5]
  >Month 6 (n=719) | 0 [0 to 4]
  >Month 9 (n=704) | 0 [0 to 5]
  >Month 12 (n=703) | 0 [0 to 5]
  Periph. lymph node enlargement (Baseline; n=729) | 0 [0 to 7]
  >Month 3 (n=726) | 0 [0 to 7]
  >Month 6 (n=719) | 0 [0 to 6]
  >Month 9 (n=704) | 0 [0 to 6]
  >Month 12 (n=703) | 0 [0 to 6]
  Lymphatic oedema, lower extrem. (Baseline; n=729) | 0 [0 to 6]
  >Month 3 (n=726) | 0 [0 to 6]
  >Month 6 (n=719) | 0 [0 to 5]
  >Month 9 (n=704) | 0 [0 to 6]
  >Month 12 (n=703) | 0 [0 to 5]

5. Secondary Outcome: Reported Adverse Events/Serious Adverse Events
Description: Adverse events (AEs) were collected during the course of the study from the first visit (Baseline) through the last visit (12 months). The number of participants experiencing a non-serious or serious adverse event or both types of events are summarized. See the Reported Adverse Event section for details.
Time Frame: Baseline to 12 months
Population: Analysis conducted in the intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Number analyzed (Participants) | 729
Participants
  Experienced a serious AE | 5
  Experienced a non-serious AE | 3
  Experienced both a serious AE and non-serious AE | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first study visit (Baseline) through the last study visit (Month 12).
Description: The adverse event population includes all enrolled participants.
Arm/Group | Advanced PCa Patients With LUTS Treated With GnRH Analogue
Serious Adverse Events (participants affected / at risk) | 6/729
Other Adverse Events (participants affected / at risk) | 0/729
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced PCa Patients With LUTS Treated With GnRH Analogue (N=729)
Renal failure (Renal and urinary disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Death (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 1 (1)
Bone pain (General disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Weight increased (Investigations) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection